CLINICAL TRIAL: NCT01156844
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel Group, Repeated-dose Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of Three Different Dosing Regimens of Inhaled Indacaterol Maleate in Patients With Persistent Asthma
Brief Title: Efficacy, Safety and Pharmacokinetics of Different Regimens of Indacaterol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAB149B2223; 2010-018481-22 (EudraCT Number)
Record Dates: First submitted 2010-06-30; First posted 2010-07-05 (Estimated); Results first posted 2011-08-17 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-07

CONDITIONS: Persistent Asthma
Keywords: Indacaterol; Asthma; Bronchodilation; Beta-agonist
MeSH Terms: conditions — Asthma | interventions — indacaterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Indacaterol 37.5 µg (twice a day) (Experimental): Indacaterol 37.5 µg twice a day (bid) inhaled via Concept1, a single dose dry powder inhaler (SDDPI), in the morning and in the evening for 16 days.
  All patients had to receive daily treatment with inhaled corticosteroid up to the maximum dose per day in a stable regimen for at least 4-weeks prior to screening and remain stable through out the study. The short acting (beta) β2-agonist (SABA) salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol
- Indacaterol 75 µg (once a day) (Experimental): Indacaterol 75 µg once a day (qd) inhaled via Concept1, a single dose dry powder inhaler (SDDPI), in the morning and Placebo to Indacaterol inhaled once daily via Concept1 in the evening for 16 days.
  All patients had to receive daily treatment with inhaled corticosteroid up to the maximum dose per day in a stable regimen for at least 4-weeks prior to screening and remain stable through out the study. The short acting (beta) β2-agonist (SABA) salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Placebo to Indacaterol
- Indacaterol 150 µg (every other day) (Experimental): Indacaterol 150 µg every other day (qod) inhaled via Concept1, a single dose dry powder inhaler (SDDPI) for a total of 16 days. Indacaterol 150 µg inhaled via Concept1, a SDDPI, in the morning and Placebo to Indacaterol inhaled via Concept1 in the evening on odd days; and Placebo to Indacaterol inhaled via Concept1 in the morning and in the evening on even days.
  All patients had to receive daily treatment with inhaled corticosteroid up to the maximum dose per day in a stable regimen for at least 4-weeks prior to screening and remain stable through out the study. The short acting (beta) β2-agonist (SABA) salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Placebo to Indacaterol
- Placebo (Placebo Comparator): Placebo to Indacaterol twice daily (bid) inhaled via Concept1, a single dose dry powder inhaler (SDDPI), in the morning and in the evening for 16 days.
  All patients had to receive daily treatment with inhaled corticosteroid up to the maximum dose per day in a stable regimen for at least 4-weeks prior to screening and remain stable through out the study. The short acting (beta) β2-agonist (SABA) salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Placebo to Indacaterol

INTERVENTIONS:
Drug: Indacaterol — Indacaterol inhaled via Concept1, a single dose dry powder inhaler (SDDPI) for 16 days. Dosage and frequency varied according to randomization scheme.
  Arms: Indacaterol 150 µg (every other day); Indacaterol 37.5 µg (twice a day); Indacaterol 75 µg (once a day)
Drug: Placebo to Indacaterol — Placebo inhaled via Concept1, a SDDPI. Frequency varied according to randomization scheme.
  Arms: Indacaterol 150 µg (every other day); Indacaterol 75 µg (once a day); Placebo

SUMMARY:
This study assessed the bronchodilator efficacy of three different regimens of indacaterol in patients with asthma

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of asthma and:
* Receiving daily treatment with inhaled corticosteroid in a regimen that has been stable for at least a month prior to screening
* FEV1 ≥50% and ≤90% of predicted normal at screening
* An increase of ≥12% and ≥200 mL in FEV1 over prebronchodilator value within 30 minutes after inhaling a total dose of albuterol/salbutamol of 360/400 MDI

Exclusion Criteria:

* Smoking history of ≥ 10 years
* Patients with a diagnosis of COPD
* Patients who have been previously intubated for a severe asthma exacerbation/ attack
* Patients who have experienced a severe asthma attack/exacerbation requiring hospitalization in the 6 months prior to screening
* Patients who have had an emergency room visit for an asthma attack/exacerbation within 6 weeks prior to screening
* Patients who have had a respiratory tract infection within 6 weeks prior to screening
* Patients with seasonal allergy whose asthma is likely to deteriorate during the study period
* Patients with Type I or uncontrolled Type II diabetes mellitus

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2010-03; Primary Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (28):
- United States (19):
  - Novartis Investigative Site, Anniston, Alabama
  - Novartis Investigative Site, Cypress, California
  - Novartis Investigative Site, Fresno, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Clearwater, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Normal, Illinois
  - Novartis Investigative Site, Lafayette, Louisiana
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Berlin, New Jersey
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigator Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Plano, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Tacoma, Washington
- France (2):
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rennes
- Novartis Investigative Site, Wiesbaden, Germany
- Jordan (2):
  - Novartis Investigative Site, Amman
  - Novartis Investigative Site, Irbid
- Novartis Investigative Site, Groningen, Netherlands
- United Kingdom (3):
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Merthyr Tydfil

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of a 21 day screening period, a 14 day run-in period and a baseline assessment day prior to the 16 day treatment period. 1 participant randomized to 75 ug Indacaterol and 1 participant randomized to Placebo did not receive study drug and were not included in the Safety set milestone.
Period: Overall Study
Arm/Group | Indacaterol 37.5 µg (Twice a Day) | Indacaterol 75 µg (Once a Day) | Indacaterol 150 µg (Every Other Day) | Placebo
Started | 48 (Randomized participants.) | 48 | 48 | 47
PD & Safety Sets: Received Study Drug | 48 (PD=Pharmacodynamic) | 47 | 48 | 46
Completed | 46 | 46 | 42 | 41
Not Completed | 2 | 2 | 6 | 6
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Abnormal test procedure result(s) | 0 | 1 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Administrative problems | 0 | 1 | 0 | 1
Not completed — Protocol deviation | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol 37.5 µg (Twice a Day) | Indacaterol 75 µg (Once a Day) | Indacaterol 150 µg (Every Other Day) | Placebo | Total
Number analyzed (Participants) | 48 | 47 | 48 | 46 | 189
Age Continuous [Mean (Standard Deviation); unit: years] — Baseline measures used the Safety Set that included all participants who received at least one dose of study drug.
  years | 37.4 (11.0) | 41.1 (14.7) | 42.0 (12.2) | 40.8 (12.7) | 40.3 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 24 | 16 | 18 | 79
  Male | 27 | 23 | 32 | 28 | 110

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Trough Forced Expiratory Volume in One Second (FEV1) After Two Weeks of Treatment
Description: Spirometry was conducted according to internationally accepted standards. Trough FEV1 values were calculated as the mean of the 23.17 hours and 23.75 hours post morning dose FEV1 measurements. Analysis of covariance model was used with baseline FEV1 as a continuous covariate.
Time Frame: Baseline to week 2
Population: Pharmacodynamic (PD) Analysis Set included all randomized participants who received at least one dose of study drug and who had evaluable PD data.
Measure: Least Squares Mean (90% Confidence Interval); unit: Liters
Arm/Group | Indacaterol 37.5 µg (Twice a Day) | Indacaterol 75 µg (Once a Day) | Indacaterol 150 µg (Every Other Day) | Placebo
Number analyzed (Participants) | 48 | 47 | 48 | 46
Liters | 0.156 [0.083 to 0.228] | 0.197 [0.125 to 0.269] | 0.199 [0.125 to 0.272] | -0.005 [-0.080 to 0.071]

2. Primary Outcome: Change From Baseline in the Forced Expiratory Volume in 1 Second Standardized (With Respect to Time) Area Under the Curve (AUC) From 0 to 24 Hours Post Dose (FEV1 AUC 0-24h) After Two Weeks of Treatment
Description: Spirometry was conducted according to internationally accepted standards. Standardized area under the curve (AUC 0-24 hours) of FEV1 measurements taken at pre-dose to 24 hours post-dose was calculated based on the trapezoidal rule and was adjusted for the area per time unit using the scheduled time of measurements for FEV1. Analysis of covariance model was used with baseline FEV1 as a continuous covariate.
Time Frame: Baseline, 0-24 hours post dose week 2
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Liters
Groups:
- Placebo: Placebo to Indacaterol twice daily (bid) inhaled via Concept1, a single dose dry powder inhaler (SDDPI), in the morning and in the evening for 16 days. All patients had to receive daily treatment with inhaled corticosteroid up to the maximum dose per day in a stable regimen for at least 4-weeks prior to screening and remain stable through out the study. The short acting (beta) β2-agonist (SABA) such as salbutamol/albuterol was available for rescue use throughout the study.
Arm/Group | Indacaterol 37.5 µg (Twice a Day) | Indacaterol 75 µg (Once a Day) | Placebo
Number analyzed (Participants) | 48 | 47 | 46
Liters | 0.196 [0.127 to 0.266] | 0.198 [0.127 to 0.269] | 0.030 [-0.044 to 0.103]

3. Primary Outcome: Change From Baseline in the Forced Expiratory Volume in 1 Second Standardized (With Respect to Time) Area Under the Curve (AUC) From 0 to 48 Hours (FEV1 AUC 0-48h) After Two Weeks of Treatment
Description: Spirometry was conducted according to internationally accepted standards. Standardized area under the curve (AUC 0-48 hours) of FEV1 measurements taken at pre-dose to 48 hours post-dose was calculated based on the trapezoidal rule and was adjusted for the area per time unit by using the scheduled time of measurements for FEV1. Analysis of covariance model was used with baseline FEV1 as a continuous covariate.
Time Frame: Baseline, 0 to 48 hours post dose week 2
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Liters
Arm/Group | Indacaterol 75 µg (Once a Day) | Indacaterol 150 µg (Every Other Day) | Placebo
Number analyzed (Participants) | 47 | 48 | 46
Liters | 0.218 [0.148 to 0.288] | 0.198 [0.135 to 0.260] | 0.059 [-0.012 to 0.129]

4. Secondary Outcome: Change From Baseline in the Forced Expiratory Volume in 1 Second Standardized (With Respect to Time) Area Under the Curve (AUC) From 0 to 12 Hours (FEV1 AUC 0-12h) After Two Weeks of Treatment
Description: Spirometry was conducted according to internationally accepted standards. Standardized area under the curve (AUC 0-12 hours) of FEV1 measurements taken at pre-dose to 12 hours post-dose was calculated based on the trapezoidal rule and was adjusted for the area per time unit by using the scheduled time of measurements for FEV1. Analysis of covariance model was used with baseline FEV1 as a continuous covariate.
Time Frame: Baseline, 0 to 12 hours post dose week 2
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Liters
Arm/Group | Indacaterol 37.5 µg (Twice a Day) | Indacaterol 75 µg (Once a Day) | Placebo
Number analyzed (Participants) | 48 | 47 | 46
Liters | 0.245 [0.170 to 0.319] | 0.243 [0.163 to 0.317] | 0.059 [-0.018 to 0.137]

ADVERSE EVENTS:
Description: Safety population.
Groups:
- Indacaterol 37.5 ug (Twice a Day): Indacaterol 37.5 µg twice a day (bid) inhaled via Concept1, a single dose dry powder inhaler (SDDPI), in the morning and in the evening for 16 days. All patients had to receive daily treatment with inhaled corticosteroid up to the maximum dose per day in a stable regimen for at least 4-weeks prior to screening and remain stable through out the study. The short acting (beta) β2-agonist (SABA) salbutamol/albuterol was available for rescue use throughout the study.
- Indacaterol 75 ug (Once a Day): Indacaterol 75 µg once a day (qd) inhaled via Concept1, a single dose dry powder inhaler (SDDPI), in the morning and Placebo to Indacaterol inhaled once daily via Concept1 in the evening for 16 days. All patients had to receive daily treatment with inhaled corticosteroid up to the maximum dose per day in a stable regimen for at least 4-weeks prior to screening and remain stable through out the study. The short acting (beta) β2-agonist (SABA) salbutamol/albuterol was available for rescue use throughout the study.
- Indacaterol 150 ug (Every Other Day): Indacaterol 150 µg every other day (qod) inhaled via Concept1, a single dose dry powder inhaler (SDDPI) for a total of 16 days. Indacaterol 150 µg inhaled via Concept1, a SDDPI, in the morning and Placebo to Indacaterol inhaled via Concept1 in the evening on odd days; and Placebo to Indacaterol inhaled via Concept1 in the morning and in the evening on even days. All patients had to receive daily treatment with inhaled corticosteroid up to the maximum dose per day in a stable regimen for at least 4-weeks prior to screening and remain stable through out the study. The short acting (beta) β2-agonist (SABA) salbutamol/albuterol was available for rescue use throughout the study.
Arm/Group | Indacaterol 37.5 ug (Twice a Day) | Indacaterol 75 ug (Once a Day) | Indacaterol 150 ug (Every Other Day) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/47 | 1/48 | 0/46
Other Adverse Events (participants affected / at risk) | 7/48 | 8/47 | 11/48 | 8/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 37.5 ug (Twice a Day) (N=48) | Indacaterol 75 ug (Once a Day) (N=47) | Indacaterol 150 ug (Every Other Day) (N=48) | Placebo (N=46)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 37.5 ug (Twice a Day) (N=48) | Indacaterol 75 ug (Once a Day) (N=47) | Indacaterol 150 ug (Every Other Day) (N=48) | Placebo (N=46)
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 1 | 1
Headache (Nervous system disorders) | 3 | 2 | 3 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.